CLINICAL TRIAL: NCT06999174
Title: Multiparametric MRI for Optimized Imaging-based Characterization and Therapy Management of Hepatocellular Carcinoma
Brief Title: Multiparametric MRI for Characterization of Hepatocellular Carcinoma
Status: Recruiting | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Emily Hoffmann, MD, University Hospital Muenster
Other Study IDs: 2025-207-f-S; University of Münster (Other Grant/Funding Number: 2025-207-f-S)
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Multiparametric MRI; TACE; SIRT
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HCC patients undergoing TACE or SIRT: Patients with hepatocellular carcinoma scheduled for TACE or SIRT, undergoing multiparametric MRI at three defined time points.
  Interventions: Diagnostic Test: Multiparametric MRI

INTERVENTIONS:
Diagnostic Test: Multiparametric MRI — Diagnostic multiparametric liver MRI, performed at three time points: before (≤14 days), 24 hours after, and 4-6 weeks after TACE or 3 months after SIRT.

SUMMARY:
This prospective observational study investigates using multiparametric magnetic resonance imaging (MRI) to improve the characterization and management of therapy for hepatocellular carcinoma (HCC). The goal is to evaluate whether advanced MRI parameters can support noninvasive diagnostic assessments and personalized treatment plans for patients with HCC. The study is being conducted at a single university center in Germany and includes adult patients with confirmed or suspected HCC. Participants will undergo standardized multiparametric MRI examinations, and the imaging data will be correlated with clinical, pathological, and therapeutic outcomes. No study-specific interventions or medications will be administered.

DETAILED DESCRIPTION:
This prospective, monocentric, observational study evaluates the clinical utility of multiparametric magnetic resonance imaging (mpMRI) in the characterization and management of hepatocellular carcinoma (HCC). The study focuses on how advanced MRI techniques-such as diffusion-weighted imaging (DWI), dynamic contrast-enhanced MRI (DCE-MRI), and quantitative mapping (T1/T2)-can provide functional insights into tumor biology.

Conducted at a German university hospital, the study investigates whether mpMRI can improve diagnostic precision and assist in therapeutic decision-making for patients undergoing locoregional treatments like transarterial chemoembolization (TACE) or selective internal radiotherapy (SIRT).

By integrating multiple MRI biomarkers, the study aims to explore correlations between imaging features and treatment response. Imaging protocols follow current clinical standards, and the study introduces no investigational agents. Radiological evaluations are performed by expert radiologists, and statistical analysis is pre-specified. The study complies with ethical and data protection standards.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Confirmed or suspected diagnosis of HCC
* Scheduled to receive TACE or SIRT as part of standard clinical care
* Eligibility for liver MRI
* Willing and able to provide written informed consent

Exclusion Criteria:

* Contraindications to MRI (e.g., pacemakers, ferromagnetic implants, severe claustrophobia)
* Known allergy or intolerance to gadolinium-based contrast agents
* Renal insufficiency with estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m²
* Pregnancy or breastfeeding
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with confirmed or suspected HCC who are scheduled for TACE or SIRT as part of routine clinical care at a tertiary academic center. Patients must be eligible for liver MRI and provide informed consent. The population includes treatment-naive as well as previously treated individuals, as long as they meet the inclusion criteria. Recruitment is non-randomized and consecutive.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of multiparametric MRI parameters with early therapy response | 4 to 6 weeks after TACE, 3 months after SIRT
  Evaluation of mpMRI features (e.g. ADC values, T1 relaxation time, enhancement patterns) in relation to early treatment response assessed 4-6 weeks after TACE or 3 months after SIRT using modified RECIST (mRECIST) criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic of Radiology, University of Münster, Münster, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will not be shared for this study. The study is observational and does not include consent for data sharing beyond internal analysis.

REFERENCES:
- [Background] Zhang C, Chen X, Wang J, Luo T. Diagnostic values of contrast-enhanced MRI and contrast-enhanced CT for evaluating the response of hepatocellular carcinoma after transarterial chemoembolisation: a meta-analysis. BMJ Open. 2024 Apr 5;14(4):e070364. doi: 10.1136/bmjopen-2022-070364. PMID 38580362
- [Background] Wang L, Yang JD, Yoo CC, Lai KKY, Braun J, McGovern DPB, Xie Y, Pandol SJ, Lu SC, Li D. Magnetic resonance imaging for characterization of hepatocellular carcinoma metabolism. Front Physiol. 2022 Dec 15;13:1056511. doi: 10.3389/fphys.2022.1056511. eCollection 2022. PMID 36589457
- [Background] Hoffmann E, Masthoff M, Kunz WG, Seidensticker M, Bobe S, Gerwing M, Berdel WE, Schliemann C, Faber C, Wildgruber M. Multiparametric MRI for characterization of the tumour microenvironment. Nat Rev Clin Oncol. 2024 Jun;21(6):428-448. doi: 10.1038/s41571-024-00891-1. Epub 2024 Apr 19. PMID 38641651